CLINICAL TRIAL: NCT04452331
Title: An Assessment of Open Access Audio of the Clinical Encounter on Veterans and Their Care
Brief Title: Assessing Open Access Audio
Acronym: OAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IIR 19-068
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The setting will be primary care and diabetes clinics, at two facilities for generalizability. To achieve aims 1 and 2, the investigators plan a randomized controlled three arm design: (1) the encounter is recorded, with provider and patient aware, and uploaded to a server the Veteran, provider, and research team can access post visit; (2) the encounter is recorded, with both parties aware, and uploaded to a server only the research team can access; and (3) the encounter is recorded, with only the patient aware, and uploaded to a server only the research team can access. Resource utilization and disease measures indicated in aims 1 and 2 will be collected in all arms.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Arm 1 is the intervention, with both provider and patient aware of the recording. It is designed to represent how OAA would be utilized in actual practice. In Arm 2 all parties are also aware of the audio recording, but this time neither gets access to the audio after the visit (although the research team does). Arm 2 is a control for isolating the effect of patient access after the visit to the audio in Arm 1. Both patient and physician are blind to whether they are in Arm 1 or 2 until after the visit. Arm 3 is a second kind of control, as the audio is again not shared with the patient. In this arm, however, the patient conceals the audio recorder, so that the provider is unaware they are being audio recorded until after the visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- OAA Intervention (Experimental): Visit recorded, both patient and provider aware, both patient and provider have access to audio post-visit
  Interventions: Other: Open Access Audio
- OAA Physician Aware Control (Sham Comparator): Visit recorded, both patient and provider aware, neither patient nor provider have access to audio post-visit
  Interventions: Other: No Access, Patient and Provider Aware of Recording
- OAA Physician Unaware Control (Placebo Comparator): Visit recorded, patient aware but provider unaware, neither patient nor provider have access to audio post-visit
  Interventions: Other: No Access, Provider Unaware of Recording

INTERVENTIONS:
Other: Open Access Audio — Patient obtains secure access to an audio recording of the medical encounter post-visit that is accessible from any internet enabled device.
  Other Names: OAA
  Arms: OAA Intervention
Other: No Access, Patient and Provider Aware of Recording — Patient does not obtain access to audio recording but both patient and provider are aware visit is being recorded.
  Other Names: OAA All Aware
  Arms: OAA Physician Aware Control
Other: No Access, Provider Unaware of Recording — Patient does not obtain access to audio recording and provider is unaware visit is being recorded.
  Other Names: OAA Provider Unaware
  Arms: OAA Physician Unaware Control

SUMMARY:
The medical encounter can be overwhelming in term of the amount of information discussed, its technical nature, and the anxiety it can generate. Easy access to a secure audio recording from any internet enabled device is an available low cost technology that allows patients to "revisit the visit" either alone or sharing with caretakers and family. It has been introduced and tested outside the VA with evidence that it increases patient recall and understanding and may even improve physician performance. Little is known, however, about whether and to what extent these effects lead to better outcomes, such as improved treatment plan adherence and chronic disease self-management. This study is a randomized controlled trial designed ascertain whether easy access to audio recordings of the medical visit improves patients perception that they understand and can manage their own care, and leads to a variety of improved outcomes, such as better blood pressure and diabetes control, and fewer emergency department visits and hospitalizations.

DETAILED DESCRIPTION:
The study aims to assess (1) the impact of an open access audio (OAA) program on two behaviors (patient activation, treatment plan adherence), and two chronic condition measures (glycosylated hemoglobin, blood pressure); (2) the impact of open access audio on provider communication and on their attention to patient contextual factors (i.e. individual Veteran's needs and circumstances relevant to planning effective care); and (3) patient, provider, and leadership perceptions of the extent to which the program is safe, not burdensome, and worthwhile at both the start and at two years into the program. A secondary analysis will descriptively measure the effect size of OAA on ED visits and hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with scheduled appointments at the participating sites: primary care and diabetes clinics at Jesse Brown VA Medical Center and the Louis Stokes Cleveland VA Medical Center

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1553 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul J. Weiner, MD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although providers are also engaged as part of the intervention, all trial enrollment, randomization, assignment, and analysis is by patient visit. It is only the patient's assignment that affects which study arm a visit with a provider falls into. Accordingly, providers are not considered "participants enrolled" for purposes of study result reporting.
Period: Overall Study
Arm/Group | OAA Intervention | OAA Physician Aware Control | OAA Physician Unaware Control
Started | 691 | 694 | 168
Completed | 691 | 694 | 168
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OAA Intervention | OAA Physician Aware Control | OAA Physician Unaware Control | Total
Number analyzed (Participants) | 691 | 694 | 168 | 1553
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.8) | 61.9 (11.6) | 61.3 (10.8) | 62.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 3 | 72
  Male | 657 | 659 | 165 | 1481
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 27 | 7 | 59
  Not Hispanic or Latino | 639 | 649 | 158 | 1446
  Unknown or Not Reported | 27 | 18 | 3 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 3 | 9
  Asian | 1 | 5 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 6 | 8 | 0 | 14
  Black or African American | 517 | 504 | 132 | 1153
  White | 140 | 151 | 24 | 315
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 25 | 22 | 8 | 55
Clinical setting [Count of Participants; unit: Participants]
  Diabetes clinic | 146 | 146 | 0 | 292
  Primary care clinic | 545 | 548 | 168 | 1261

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: This outcome tests the hypothesis that blood pressure control improves in patients with blood pressure > 140/90 when they have access to an audio recording of their visit with their provider regarding blood pressure management compared to those who do not. An improvement in blood pressure is defined as a reduction of 10 or more mmHg in either the systolic or diastolic blood pressure.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 691 | 694
mmHg
  Systolic | 131.6 [129.9 to 133.3] | 131.8 [130.1 to 133.5]
  Diastolic | 78.2 [77.3 to 79.2] | 79.5 [78.6 to 80.5]
Statistical Analysis 1: Comparison: OAA Intervention vs OAA Physician Aware Control; Diastolic BP; Test type: Superiority; p = 0.06, Regression, Linear; Adjusted for clinical site
Statistical Analysis 2: Comparison: OAA Intervention vs OAA Physician Aware Control; Systolic BP; Test type: Superiority; p = 0.90, Regression, Linear

2. Primary Outcome: Glycosylated Hemoglobin (HgB A1c)
Description: This outcome tests the hypothesis that HgB A1c improves in patients with Hgb A1c > 7 when they have access to an audio recording of their discussion with their provider regarding diabetes management compared to when they do no. An improvement is defined as a decrease of 1% or more.
Time Frame: 4-6 months
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 691 | 694
percent | 6.95 [6.79 to 7.12] | 6.83 [6.66 to 7.00]

3. Primary Outcome: Return Visit Adherence (RVA)
Description: This outcome tests the hypothesis that return visit adherence (RVA) improves in patients with non-adherence when they have access to an audio recording of their discussion with their provider. The outcome is the predicted proportion of visits scheduled between the time of the index visit and the end of the study that the patient attends (adjusted for clinic). For example, a value of 0.73 means that, adjusted for clinic, a patient in the given arm attends 73% of visits scheduled between their index visit and the study end date.
Time Frame: From index visit to end of study data collection, an average of 512 days
Measure: Number (95% Confidence Interval); unit: Proportion of future visits attended
Units Other Than Participants: scheduled visits
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 691 | 694
Number analyzed (scheduled visits) | 12704 | 12685
Proportion of future visits attended | 0.733 [0.72 to 0.75] | 0.732 [0.72 to 0.75]
Statistical Analysis 1: Comparison: OAA Intervention vs OAA Physician Aware Control; Test type: Superiority; p = .29, Regression, Linear

4. Primary Outcome: Prescription Refill Rate (Probability That Proportion Days Covered >= 80%)
Description: This outcome tests the hypothesis that prescription adherence improves in patients when they have access to an audio recording of their discussion with their provider compared to when they do not. Adherence is defined as having at least 80% proportion days covered (PDF). PDC is the total number of days covered by refills in a measurement period divided by the number of days between the first fill and the end of the measurement period. Non-adherence is defined as a PDC<80% during the 6 months prior to the audio recorded visit. The outcome is the probability that a patient's PDC is at least 80% following their participation, adjusted for clinic.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Probability of >=80% PDC
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 691 | 694
Probability of >=80% PDC | 0.05 [0.04 to 0.06] | 0.04 [0.03 to 0.05]
Statistical Analysis 1: Comparison: OAA Intervention vs OAA Physician Aware Control; Test type: Superiority; p = .10, Regression, Logistic

5. Primary Outcome: Patient Activation Measure (PAM)
Description: This outcome tests the hypothesis that patient activation is higher in patients when they have access to an audio recording of their visit with their provider compared to when they do not. Patients are called by phone post visit to answer PAM 10, a 10 item questionnaire with a 5 point Likert response that scores their perceived knowledge, skills, and confident in their capacity to follow their treatment plan with scores from 0-100. A higher score indicates higher patient activation.
Time Frame: 2 weeks
Population: Random samples from arms 1 and 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 295 | 301
score on a scale | 9.44 [9.26 to 9.62] | 9.54 [9.37 to 9.71]
Statistical Analysis 1: Comparison: OAA Intervention vs OAA Physician Aware Control; Test type: Superiority; p = 0.44, Regression, Linear

6. Primary Outcome: SEGUE Framework for Evaluating and Scoring Communication Behavior.
Description: This outcome tests the hypothesis that physicians communicate more effectively when they are aware the visit is being recorded for the patient to when they are not. Communication behavior will be rated off the audio recording by a research assistant utilizing the SEGUE checklist. Outcome measure is total proportion achieved score on 32 item SEGUE instrument, ranging from 0 to 1 with a higher score indicating more effective communication.
Time Frame: Recorded visit
Population: Arm 2 random subsample compared with Arm 3, excluding visits with no recordings due to recorder failure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OAA Physician Aware Control | OAA Physician Unaware Control
Number analyzed (Participants) | 158 | 158
score on a scale | 0.85 [0.83 to 0.87] | 0.82 [0.80 to 0.83]
Statistical Analysis 1: Comparison: OAA Physician Aware Control vs OAA Physician Unaware Control; Test type: Superiority; p = 0.01, Regression, Linear

7. Primary Outcome: Contextualization of Care
Description: This outcome tests the hypothesis that physicians are more likely to contextualize the care plan when they are aware the visit is being recorded for the patient to when they are not. Contextualization of care will be rated off of the audio recording by a research assistant trained in Content Coding for Contextualization of Care (4C Coding), which determines each contextual red flag audible during the visit, whether the physician probed each red flag, each contextual factor identified by physician probe, and whether the physician addressed the contextual factor in the care plan. Outcome measure is the predicted probability of an encounter in which the care plan was contextualized (either the physician found no contextual factors present after investigating red flags, or physician found a contextual factor(s) and incorporated them into the plan), adjusted for clinic.
Time Frame: Recorded visit
Population: Arm 2 random subsample vs. Arm 3, excluding visits with recorder failure or on phone
Measure: Number (95% Confidence Interval); unit: Predicted probability of contextual plan
Arm/Group | OAA Physician Aware Control | OAA Physician Unaware Control
Number analyzed (Participants) | 158 | 160
Predicted probability of contextual plan | 0.51 [0.45 to 0.56] | 0.41 [0.35 to 0.47]
Statistical Analysis 1: Comparison: OAA Physician Aware Control vs OAA Physician Unaware Control; Test type: Superiority; p = 0.01, Regression, Logistic

8. Secondary Outcome: Emergency Department Utilization
Description: This outcome tests the hypothesis that emergency department visit rates are lower following encounters in which patients have access to an audio recording of their visit with their provider compared to when they do not. Outcome measure is the average number of ED visits made by the patient in the 6 months following the audio recorded visit, adjusted for clinic.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: ED visits
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 691 | 694
ED visits | 1.03 [0.88 to 1.19] | 0.96 [0.83 to 1.12]
Statistical Analysis 1: Comparison: OAA Intervention vs OAA Physician Aware Control; Test type: Superiority; p = 0.54, Regression, negative binomial

9. Secondary Outcome: Hospital Admission Rate
Description: This outcome tests the hypothesis that inpatient admission rates are lower following encounters in which patients have access to an audio recording of their visit with their provider compared to when they do not. Outcome measure is the average number of inpatient hospital admissions of the patient (of any duration) during the 6 month period following the audio recorded visit.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Hospital admissions
Arm/Group | OAA Intervention | OAA Physician Aware Control
Number analyzed (Participants) | 691 | 694
Hospital admissions | 0.26 [0.21 to 0.33] | 0.28 [0.22 to 0.35]
Statistical Analysis 1: Comparison: OAA Intervention vs OAA Physician Aware Control; Test type: Superiority; p = 0.74, Regression, negative binomial

10. Secondary Outcome: Glycated Hemoglobin (Access vs. Non-access)
Description: Comparison of HgA1c among Arm 1 patients who did and did not access their visit recording
Time Frame: Six month
Measure: Mean (95% Confidence Interval); unit: percent
Groups:
- OAA Intervention + Accessed: Visit recorded, both patient and provider aware, both patient and provider have access to audio post-visit, patient accesses the recording.
  Open Access Audio: Patient obtains secure access to an audio recording of the medical encounter post-visit that is accessible from any internet enabled device.
- OAA Intervention + Not Accessed: Visit recorded, both patient and provider aware, both patient and provider have access to audio post-visit, patient does not access the recording.
  Open Access Audio: Patient obtains secure access to an audio recording of the medical encounter post-visit that is accessible from any internet enabled device.
Arm/Group | OAA Intervention + Accessed | OAA Intervention + Not Accessed | OAA Physician Aware Control
Number analyzed (Participants) | 153 | 520 | 694
percent | 6.53 [6.20 to 6.85] | 6.95 [6.78 to 7.12] | 6.73 [6.58 to 6.88]
Statistical Analysis 1: Comparison: OAA Intervention + Accessed vs OAA Intervention + Not Accessed; Test type: Superiority; p = 0.03, Regression, Linear
Statistical Analysis 2: Comparison: OAA Intervention + Not Accessed vs OAA Physician Aware Control; Test type: Superiority; p = 0.06, Regression, Linear

11. Secondary Outcome: ED Visit Rate (Access vs. Non-access)
Description: Comparison of ED visit rate among Arm 1 patients who did and did not access their visit recording. The ED visit rate is the number of emergency department visits in the 6 months following the patient's recorded visit, adjusted for clinic.
Time Frame: Six month
Measure: Mean (95% Confidence Interval); unit: ED visits
Arm/Group | OAA Intervention + Accessed | OAA Intervention + Not Accessed | OAA Physician Aware Control
Number analyzed (Participants) | 153 | 520 | 694
ED visits | 0.69 [0.57 to 0.84] | 1.05 [0.97 to 1.14] | 0.93 [0.86 to 1.00]
Statistical Analysis 1: Comparison: OAA Intervention + Accessed vs OAA Intervention + Not Accessed; Test type: Superiority; p < 0.001, Regression, negative binomial
Statistical Analysis 2: Comparison: OAA Intervention + Not Accessed vs OAA Physician Aware Control; Test type: Superiority; p = 0.03, Regression, negative binomial

12. Secondary Outcome: Return Visit Attendance (Access vs. Non-access)
Description: Comparison of RVA among Arm 1 patients who did and did not access their visit recording. The outcome is the predicted proportion of visits scheduled between the time of the index visit and the end of the study that the patient attends (adjusted for clinic). For example, a value of 0.73 means that, adjusted for clinic, a patient in the given arm attends 73% of visits scheduled between their index visit and the study end date.
Time Frame: From recorded visit to study end date, an average of 512 days
Population: Patients in OAA intervention arm (accessed and not access) exclude 11 patients who did not have the opportunity to access a recording due to recorder failure.
Measure: Number (95% Confidence Interval); unit: Proportion of return visits attended
Arm/Group | OAA Intervention + Accessed | OAA Intervention + Not Accessed | OAA Physician Aware Control
Number analyzed (Participants) | 153 | 527 | 694
Proportion of return visits attended | 0.78 [0.75 to 0.82] | 0.71 [0.70 to 0.73] | 0.73 [0.72 to 0.75]
Statistical Analysis 1: Comparison: OAA Intervention + Accessed vs OAA Intervention + Not Accessed; Test type: Superiority; p < 0.001, Regression, poisson
Statistical Analysis 2: Comparison: OAA Intervention + Not Accessed vs OAA Physician Aware Control; Test type: Superiority; p = 0.08, Regression, poisson

13. Secondary Outcome: Probability That Proportion of Days Covered by Prescription >= 80% (Access vs. Non-access)
Description: Comparison of probability of prescription refill adherence (PDC>=80%) among Arm 1 patients who did and did not access their visit recording. Adherence is defined as having at least 80% proportion days covered (PDF). PDC is the total number of days covered by refills in a measurement period divided by the number of days between the first fill and the end of the measurement period. Non-adherence is defined as a PDC<80% during the 6 months prior to the audio recorded visit. The outcome is the probability that a patient's PDC is at least 80% following their participation, adjusted for clinic.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Probability of at least 80% PDC
Arm/Group | OAA Intervention + Accessed | OAA Intervention + Not Accessed | OAA Physician Aware Control
Number analyzed (Participants) | 153 | 520 | 694
Probability of at least 80% PDC | 0.09 [0.06 to 0.13] | 0.04 [0.03 to 0.05] | 0.05 [0.03 to 0.05]
Statistical Analysis 1: Comparison: OAA Intervention + Accessed vs OAA Intervention + Not Accessed; Test type: Superiority; p < .001, Mixed Models Analysis; Mixed effects logistic regression including random effect of visit, to incorporate clustering of prescriptions within visits
Statistical Analysis 2: Comparison: OAA Intervention + Not Accessed vs OAA Physician Aware Control; Test type: Superiority; p = 0.98, Mixed Models Analysis; [statistical method as in outcome 13, analysis 1]

14. Secondary Outcome: Blood Pressure (Access vs. Non-access)
Description: Comparison of blood pressure among Arm 1 patients who did and did not access their visit recording
Time Frame: Six month
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | OAA Intervention + Accessed | OAA Intervention + Not Accessed | OAA Physician Aware Control
Number analyzed (Participants) | 153 | 520 | 694
mmHg
  Systolic | 130.7 [127.8 to 133.7] | 133.0 [131.3 to 134.6] | 132.7 [131.3 to 134.1]
  Diastolic | 78.0 [76.3 to 79.6] | 79.5 [78.6 to 80.4] | 80.5 [79.7 to 81.3]
Statistical Analysis 1: Comparison: OAA Intervention + Accessed vs OAA Intervention + Not Accessed; Systolic BP; Test type: Superiority; p = 0.20, Regression, Linear
Statistical Analysis 2: Comparison: OAA Intervention + Not Accessed vs OAA Physician Aware Control; Systolic BP; Test type: Superiority; p = 0.82, Regression, Linear
Statistical Analysis 3: Comparison: OAA Intervention + Accessed vs OAA Intervention + Not Accessed; Diastolic BP; Test type: Superiority; p = 0.12, Regression, Linear
Statistical Analysis 4: Comparison: OAA Intervention + Not Accessed vs OAA Physician Aware Control; Diastolic BP; Test type: Superiority; p = 0.10, Regression, Linear

ADVERSE EVENTS:
Time Frame: At recorded trial visit only
Arm/Group | OAA Intervention | OAA Physician Aware Control | OAA Physician Unaware Control
All-Cause Mortality (participants affected / at risk) | 0/691 | 0/694 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/691 | 0/694 | 0/168
Other Adverse Events (participants affected / at risk) | 0/691 | 0/694 | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04452331/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT04452331/ICF_000.pdf